CLINICAL TRIAL: NCT07199426
Title: The Effect of Physical-Cognitive Training on Balance and Falls in Older Adults
Brief Title: Effect of Physical-Cognitive Training in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gözde Baş Başer, MSc, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-FTR-GBB-01
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Older Adults, Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical-Cognitive Training Group (Experimental): Blazepod-based physical-cognitive training (8 weeks, 3 sessions/week)
  Interventions: Other: Physical-Cognitive Training
- Conventional Balance Training Group (Active Comparator): Conventional balance training (8 weeks, 3 sessions/week)
  Interventions: Other: Conventional Balance Training

INTERVENTIONS:
Other: Physical-Cognitive Training — Participants will receive an 8-week physical-cognitive training program using the Blazepod device, consisting of exercises targeting both balance and cognitive skills. Sessions will be conducted three times per week, each lasting one hour.
  Arms: Physical-Cognitive Training Group
Other: Conventional Balance Training — Participants will receive an 8-week conventional balance training program. Sessions will be conducted three times per week, each lasting one hour.
  Arms: Conventional Balance Training Group

SUMMARY:
The study compares the impact of physical-cognitive exercises using Blazepod device versus conventional balance training on multiple outcomes in older adults aged 70 and above. Participants receive an 8-week intervention, three sessions per week for both groups. Outcome measures include balance assessments, fear of falling scales, activity of daily living performance, sleep quality questionnaires, reaction time tests, and cognitive assessments. The study aims to determine whether physical-cognitive training provides additional benefits compared to conventional balance exercises.

DETAILED DESCRIPTION:
Worldwide and in Turkey, increasing life expectancy and the growth of the elderly population are associated with rising care, health, and social needs among older adults. Aging induces physiological changes that lead to declines in both physical and cognitive capacities. Recently, non-pharmacological interventions have gained importance over pharmacological treatments to improve function and avoid polypharmacy. Strength, aerobic, and balance exercises have been shown to induce structural and functional brain adaptations, increase BDNF secretion, and positively influence both physical and cognitive domains.

Systematic reviews suggest that combining cognitive training with physical exercises produces greater cognitive benefits than physical exercises alone. Conventional balance training programs for healthy older adults are widely reported in the literature, often including static and dynamic exercises performed with eyes open or closed. These exercises improve balance, reduce falls, and enhance quality of life.

However, traditional balance exercises may have limitations due to the absence of visual stimuli or reduced environmental challenges, which can limit their transfer to real-life daily activities. Recently, combined physical-cognitive training programs have gained attention.

The Blazepod system, controlled via a smartphone application, provides visual stimuli through LED lights to train reaction time and skill acquisition, while engaging both physical and cognitive processes simultaneously. Unlike conventional programs, Blazepod allows unpredictable sequences of stimuli, requiring participants to respond in real time, thus activating both physical and cognitive skills.

The aim of this study is to investigate the effects of simultaneous physical-cognitive training using Blazepod and conventional balance exercises on cognitive function, balance, daily activity performance, fall risk, and sleep quality in older adults.

This study will include two groups of participants aged 70 years and older with a Mini-Mental State Examination (MMSE) score of 24 or higher who are able to walk independently. Each group will include 17 participants, for a total of 34 participants. Both groups will participate in an 8-week intervention, three sessions per week.

In the physical-cognitive exercise group, each session will begin with a warm-up period including strengthening and mobilization exercises, followed by a Blazepod-based exercise program designed to simultaneously train balance and cognitive skills. Each session will conclude with a cool-down program including stretching and breathing exercises.

In the balance exercise group, sessions will follow the same structure: after warm-up exercises, participants will perform conventional balance exercises, followed by the same cool-down program as the physical-cognitive group.

ELIGIBILITY:
Inclusion Criteria:

* Score of 24 or higher on the Standardized Mini-Mental State Examination (MMSE)
* Ability to walk independently without assistance
* Willingness to provide written informed consent

Exclusion Criteria:

* Participation in another clinical study during the study period
* Presence of neurological or psychiatric diagnoses
* Conditions that impair walking or mobility
* Uncontrolled hypertension or cardiovascular disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Standartized Mini Mental Test | From enrollment to the end of treatment at 8 weeks
  It is a test used to assess cognitive impairment and changes, scored out of 30 points, with scores below 24 indicating potential dementia.
Montreal Cognitive Assessment | From enrollment to the end of treatment at 8 weeks
  A brief cognitive screening tool evaluating memory, attention, language, visuospatial skills, and executive function. Scores below 26 suggest possible cognitive impairment.
Fullerton Advanced Balance Scale | From enrollment to the end of treatment at 8 weeks
  A clinical balance assessment consisting of 10 tasks that test static and dynamic balance, anticipatory postural adjustments, and sensory integration. Total score is changed 0-40 and higher scores indicated better balance.
Functional Reach Test | From enrollment to the end of treatment at 8 weeks
  Assesses the maximal distance a person can reach forward beyond arm's length while maintaining a fixed base of support. Measures dynamic balance and risk of falling.
Timed Up and Go Test | From enrollment to the end of treatment at 8 weeks
  Measures the time taken to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Evaluates mobility, balance and fall risk.
Modified Falls Efficacy Scale | From enrollment to the end of treatment at 8 weeks
  Assesses fear of falling and confidence in performing daily activities. A self-reported questionnaire measuring perceived confidence in avoiding falls during various daily activities.
Deary-Liewald Reaction Time Task | From enrollment to the end of treatment at 8 weeks
  Evaluates simple and choice reaction time. A computerized test measuring the speed of cognitive-motor responses to visual stimuli.

SECONDARY OUTCOMES:
Katz Index of Independence in Activities of Daily Living | From enrollment to the end of treatment at 8 weeks
  Evaluates independence in six daily activities: bathing, dressing, toileting, transferring, continence, and feeding. Higher scores indicate greater independence.
Lawton Instrumental Activities of Daily Living Scale | From enrollment to the end of treatment at 8 weeks
  Assesses more complex daily living skills. Measures ability to perform tasks such as using the telephone, shopping, preparing meals, housekeeping, laundry, transportation, medication management, and handling finances. Higher scores indicate greater functional ability, and score is between 0-17.
Pittsburgh Sleep Quality Index | From enrollment to the end of treatment at 8 weeks
  Assess sleep quality and disturbances. A self-reported questionnaire evaluating sleep quality over the past month, including components such as sleep duration, latency, efficiency, disturbances, and daytime dysfunction. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No